CLINICAL TRIAL: NCT03697187
Title: An Observational Patient Registry to Evaluate the Real-world Safety of Ruconest® (C1 Esterase Inhibitor [Recombinant]) for the Treatment of Hereditary Angioedema
Brief Title: Patient Registry to Evaluate the Real-world Safety of Ruconest®
Status: Completed | Type: Observational
Sponsor: Pharming Technologies B.V. (Industry)
Collaborators: US Hereditary Angioedema Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: C1 1414
Record Dates: First submitted 2018-08-09; First posted 2018-10-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2020-03

CONDITIONS: Hereditary Angioedema
Keywords: Hereditary Angioedema; HAE; Ruconest; rhC1INH; Registry; Pharming
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — conestat alfa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hereditary Angioedema: Patients with Hereditary Angioedema who are receiving treatment with Ruconest (rhC1INH).
  Interventions: Drug: rhC1INH

INTERVENTIONS:
Drug: rhC1INH — Recombinant human C1 inhibitor
  Other Names: Ruconest

SUMMARY:
This is a prospective, real-world, observational patient registry for patients with HAE who are receiving treatment with Ruconest for HAE.

DETAILED DESCRIPTION:
See below.

ELIGIBILITY:
Inclusion Criteria:

1. Patient provides informed consent as documented on the Institutional Review Board (IRB) approved informed consent document (ICF). For patients aged between 13 and 17 years old, the method of consent with or without assent will be determined by the IRB.
2. Patient is male or female and at least 13 years of age at the time of providing consent / assent.
3. Patient has been prescribed Ruconest for HAE.

Exclusion Criteria:

1. Patient is receiving HAE therapy as part of a clinical trial.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients will be 13 years of age and older, have a current diagnosis of HAE for which they have been prescribed and are currently being treated with Ruconest.
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Safety analysis will consist of AEs reported per patient for up to 30 days after each single or repeated dose of Ruconest. | 3 years
  In addition, extent of exposure to Ruconest and concomitant medications taken for HAE will be summarized. Concomitant medications will be limited to those specifically indicated for treatment AEs or treatment of symptoms of HAE, for example C1-inhibitors, epinephrine, IV fluids, etc. AEs will be summarized as incidence per 10,000 person-days where each patient counts only once for multiple events of the same System Organ Class and preferred terms within the 30-day evaluation period. The person-time duration for each AE for each patient is the time period (in days) between the dose of Ruconest and AE onset.

SECONDARY OUTCOMES:
AEs occurring during pregnancy or lactation and for breastfed infants will be summarized separately using the same methods as described in the primary outcome measure. | 3 years
  Any pregnant woman who treats with Ruconest while on the Registry will be followed up to twelve weeks post-delivery or termination. Those treated with Ruconest while actively nursing will be followed until end of lactation.

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Relan, MD, Study Director — Pharming Technologies BV
Locations (1):
- The US Hereditary Angioedema Association, Fairfax, Virginia, United States